CLINICAL TRIAL: NCT07225452
Title: Liquid Biopsy Using Exosomal miRNA for Intrahepatic Cholangiocarcinoma Detection
Brief Title: An Exosomal miRNA-based Liquid Biopsy for ICC Detection
Acronym: LUMIC
Status: Recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23228/LUMIC
Record Dates: First submitted 2025-11-04; First posted 2025-11-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Intrahepatic Cholangiocarcinoma (Icc)
Keywords: ICC; Exosome; microRNA; miRNA; liquid biopsy; liver cancer
MeSH Terms: conditions — Cholangiocarcinoma; Cirrhosis, Familial, with Pulmonary Hypertension; Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Intrahepatic Cholangiocarcinoma (Discovery, Small RNA-seq): Serum and plasma samples from patients with histologically confirmed ICC will be analyzed using small RNA sequencing to identify circulating miRNAs specifically upregulated in ICC. These miRNAs will serve as candidates for downstream validation.
  Interventions: Diagnostic Test: Small RNA sequencing
- Non-disease Control (Discovery, Small RNA-seq): Serum and plasma samples from individuals without malignant or inflammatory liver diseases (benign or healthy controls) will be analyzed in parallel by small RNA sequencing to identify miRNAs differentially expressed between ICC and non-disease controls.
  Interventions: Diagnostic Test: Small RNA sequencing
- Intrahepatic Cholangiocarcinoma (Training): Patients with histologically confirmed ICC whose pre-treatment serum or plasma samples will be used to construct and optimize the exo-miRNA diagnostic panel based on discovery-phase candidates.
  Interventions: Diagnostic Test: LUMIC assay
- Non-disease Control (Training): Individuals without malignant or inflammatory liver diseases (benign or healthy controls) whose serum/plasma samples will serve as controls to establish baseline miRNA expression and diagnostic thresholds.
  Interventions: Diagnostic Test: LUMIC assay
- Intrahepatic Cholangiocarcinoma (Validation): Independent ICC cohort used for external validation of the LUMIC assay to confirm diagnostic performance and reproducibility.
  Interventions: Diagnostic Test: LUMIC assay
- Non-disease Control (Validation): Individuals without malignant or inflammatory liver diseases (benign or healthy controls) whose serum/plasma samples will be used for validation of specificity and model robustness.
  Interventions: Diagnostic Test: LUMIC assay

INTERVENTIONS:
Diagnostic Test: Small RNA sequencing — Small RNA sequencing of serum/plasma RNA to identify ICC-specific upregulated miRNAs
  Groups: Intrahepatic Cholangiocarcinoma (Discovery, Small RNA-seq); Non-disease Control (Discovery, Small RNA-seq)
Diagnostic Test: LUMIC assay — RT-qPCR validation of selected miRNAs
  Groups: Intrahepatic Cholangiocarcinoma (Training); Intrahepatic Cholangiocarcinoma (Validation); Non-disease Control (Training); Non-disease Control (Validation)

SUMMARY:
Intrahepatic cholangiocarcinoma (ICC) is a malignant liver tumor with poor prognosis and limited curative treatment options. Early and accurate detection remains an unmet clinical need.

The LUMIC study aims to develop a non-invasive liquid biopsy platform based on both exosomal microRNAs (exo-miRNAs) to detect intrahepatic cholangiocarcinoma with high sensitivity and specificity.

DETAILED DESCRIPTION:
Intrahepatic cholangiocarcinoma (ICC) is the second most common primary liver malignancy after hepatocellular carcinoma, accounting for approximately 10-15% of all primary liver cancers. Despite improvements in surgical techniques and imaging modalities, ICC is often diagnosed at advanced stages, resulting in dismal outcomes with a 5-year overall survival rate of 25-30%.

Traditional imaging approaches such as CT and MRI have limited sensitivity for detecting early or small ICC lesions. Blood-based biomarkers, including CA19-9, also lack adequate specificity.

Recent advances in liquid biopsy have demonstrated that exosomal microRNAs (exo-miRNAs) can serve as promising, minimally invasive biomarkers reflecting tumor biology and microenvironmental changes.

The LUMIC study (Liquid biopsy Using exosomal miRNA for Intrahepatic Cholangiocarcinoma detection) aims to identify and validate miRNA signatures capable of distinguishing ICC from benign biliary or non-cancerous liver conditions.

Blood samples are collected before treatment, and exo-miRNA expression profiles are analyzed using RT-qPCR and bioinformatic pipelines. Diagnostic performance (AUC, sensitivity, specificity) will be evaluated through training and validation cohorts.

This study provides a foundation for integrating liquid biopsy-based diagnostics into ICC clinical workflows to enable earlier detection and improved treatment stratification.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically confirmed intrahepatic cholangiocarcinoma
* Availability of pre-treatment plasma sample
* Informed consent provided

Exclusion Criteria:

* Extrahepatic cholangiocarcinoma
* History of other malignancy within 5 years
* Active infection, autoimmune disease, or pregnancy
* Inadequate clinical data or poor sample quality

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed with intrahepatic cholangiocarcinoma and control participants (non-cancer or benign biliary disease) with available pre-treatment plasma samples.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | Through study completion (~1 year)
  The proportion of true positive ICC cases correctly identified by the LUMIC assay.

SECONDARY OUTCOMES:
Specificity | Through study completion (~1 year)
  The proportion of true negative cases correctly classified as non-ICC.
Diagnostic accuracy (AUC) | Through study completion (~1 year)
  The overall discriminative ability of the exo-miRNA panel for ICC detection.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Goel, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

IPD SHARING:
Plan to Share IPD: No
Data collected for the study will be made available to others, including de-identified participant data, at publication, via a signed data access agreement and at the discretion of the investigators' approval of the proposed use of such data

REFERENCES:
- [Background] Li J, Bao H, Huang Z, Liang Z, Lin N, Ni C, Xu Y. Non-Coding RNA in Cholangiocarcinoma: An Update. Front Biosci (Landmark Ed). 2023 Aug 18;28(8):173. doi: 10.31083/j.fbl2808173. PMID 37664914
- [Background] Sato K, Glaser S, Alvaro D, Meng F, Francis H, Alpini G. Cholangiocarcinoma: novel therapeutic targets. Expert Opin Ther Targets. 2020 Apr;24(4):345-357. doi: 10.1080/14728222.2020.1733528. Epub 2020 Feb 26. PMID 32077341
- [Background] Luo C, Xin H, Zhou Z, Hu Z, Sun R, Yao N, Sun Q, Borjigin U, Wu X, Fan J, Huang X, Zhou S, Zhou J. Tumor-derived exosomes induce immunosuppressive macrophages to foster intrahepatic cholangiocarcinoma progression. Hepatology. 2022 Oct;76(4):982-999. doi: 10.1002/hep.32387. Epub 2022 Feb 28. PMID 35106794
- [Background] Li Z, Shen J, Chan MT, Wu WK. The role of microRNAs in intrahepatic cholangiocarcinoma. J Cell Mol Med. 2017 Jan;21(1):177-184. doi: 10.1111/jcmm.12951. Epub 2016 Sep 13. PMID 27619971
- [Background] Wada Y, Shimada M, Morine Y, Ikemoto T, Saito Y, Baba H, Mori M, Goel A. A blood-based noninvasive miRNA signature for predicting survival outcomes in patients with intrahepatic cholangiocarcinoma. Br J Cancer. 2022 May;126(8):1196-1204. doi: 10.1038/s41416-022-01710-z. Epub 2022 Jan 25. PMID 35079106
- [Background] Liu L, Shi Y, Zhang P, Zhang X. Integration analysis of miRNA-mRNA expression exploring their potential roles in intrahepatic cholangiocarcinoma. Sci Rep. 2023 May 24;13(1):8362. doi: 10.1038/s41598-023-35288-0. PMID 37225858
- [Background] European Association for the Study of the Liver. EASL-ILCA Clinical Practice Guidelines on the management of intrahepatic cholangiocarcinoma. J Hepatol. 2023 Jul;79(1):181-208. doi: 10.1016/j.jhep.2023.03.010. Epub 2023 Apr 20. PMID 37084797
- [Background] Bridgewater J, Galle PR, Khan SA, Llovet JM, Park JW, Patel T, Pawlik TM, Gores GJ. Guidelines for the diagnosis and management of intrahepatic cholangiocarcinoma. J Hepatol. 2014 Jun;60(6):1268-89. doi: 10.1016/j.jhep.2014.01.021. Epub 2014 Mar 27. No abstract available. PMID 24681130
- [Background] Moris D, Palta M, Kim C, Allen PJ, Morse MA, Lidsky ME. Advances in the treatment of intrahepatic cholangiocarcinoma: An overview of the current and future therapeutic landscape for clinicians. CA Cancer J Clin. 2023 Mar;73(2):198-222. doi: 10.3322/caac.21759. Epub 2022 Oct 19. PMID 36260350
- [Background] Tovar-Camargo OA, Toden S, Goel A. Exosomal microRNA Biomarkers: Emerging Frontiers in Colorectal and Other Human Cancers. Expert Rev Mol Diagn. 2016;16(5):553-67. doi: 10.1586/14737159.2016.1156535. Epub 2016 Mar 16. PMID 26892862
- [Background] Sui S, Xu C, Kanda M, Okugawa Y, Toiyama Y, Park JO, Hur H, Kim SC, Taketomi A, Kodera Y, Cheng X, Li M, Goel A. Exosomal Liquid Biopsy for the Early Detection of Gastric Cancer: The DESTINEX Multicenter Study. JAMA Surg. 2025 Sep 1;160(9):973-982. doi: 10.1001/jamasurg.2025.2493. PMID 40737022
- [Background] Nakamura K, Zhu Z, Roy S, Jun E, Han H, Munoz RM, Nishiwada S, Sharma G, Cridebring D, Zenhausern F, Kim S, Roe DJ, Darabi S, Han IW, Evans DB, Yamada S, Demeure MJ, Becerra C, Celinski SA, Borazanci E, Tsai S, Kodera Y, Park JO, Bolton JS, Wang X, Kim SC, Von Hoff D, Goel A. An Exosome-based Transcriptomic Signature for Noninvasive, Early Detection of Patients With Pancreatic Ductal Adenocarcinoma: A Multicenter Cohort Study. Gastroenterology. 2022 Nov;163(5):1252-1266.e2. doi: 10.1053/j.gastro.2022.06.090. Epub 2022 Jul 16. PMID 35850192